CLINICAL TRIAL: NCT01531530
Title: Safety, Clinical Tolerance, and Immunogenicity of CVD 1208S, a Delta guaBA, Delta Sen, Delta Set, Live, Oral Shigella Flexneri 2a Vaccine Manufactured Using cGMP
Brief Title: Safety and Efficacy Study of CVD 1208S, a Live, Attenuated Oral Vaccine to Prevent Shigella Infection Using cGMP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: PATH (Other)
Responsible Party: Principal Investigator, Karen Kotloff, Professor of Pediatrics, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HP-00049727; Shigella CVD 28000 (Other: Center for Vaccine Development (CVD), UMB)
Record Dates: First submitted 2011-10-26; First posted 2012-02-13 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Shigella
Keywords: Shigella; Vaccine; Mucosal immunity
MeSH Terms: conditions — Dysentery, Bacillary | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccine-recipients (Experimental)
  Interventions: Biological: CVD 1208S, a Shigella flexneri 2a live, oral vaccine
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: CVD 1208S, a Shigella flexneri 2a live, oral vaccine — The vaccine is mixed with salt water and given by mouth.
  Arms: Vaccine-recipients
Other: Placebo — Corn starch and baking soda are mixed with salt water and given by mouth.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether CVD 1208S (a live, attenuated, oral vaccine) is safe and effective in the prevention of Shigella infection.

DETAILED DESCRIPTION:
There are two purposes for conducting this Vaccine Study to evaluate an experimental vaccine called CVD 1208S (Center for Vaccine Development 1208S): 1) to learn whether CVD 1208S causes side effects, and 2) to learn whether the CVD 1208S gives people immunity to Shigella.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45 years, inclusive.
* Good general health
* Expressed interest and availability to fulfill study requirements
* Informed, written consent.
* Agrees to indefinite storage of unused clinical specimens at the CVD for use in future research
* Agrees not to participate in another investigational vaccine or drug trial during the study
* Has no childbearing potential or agrees to abstain from becoming pregnant from the day of screening (at least 14 days before vaccination) until 6 weeks after the final vaccination by using birth control
* Agrees not to donate blood to a blood bank for 12 months after receiving the vaccine.

Exclusion Criteria:

* An acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses.
* Any current illness requiring daily medication (vitamins, birth control pills, nasal or topical medications, allowed);
* Blood in stool on >2 occasions (other than small amounts from straining) in past 12 months;
* Recurrent diarrhea (>5 episodes in past 6 months, each lasting 3 days or more).
* Immunosuppression
* Long term (greater than 2 weeks) use of oral or injected steroids, or high-dose inhaled steroids (>800 micrograms/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (Nasal and topical steroids are allowed).
* History of abdominal surgery
* Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* Known allergy or intolerance to ciprofloxacin, trimethoprim/sulfamethoxazole (or other sulfa antibiotic), ampicillin (for women) or corn.
* History of shigellosis or Shigella vaccination or challenge or a laboratory worker with known exposure to Shigella.
* Anticipates any of the following during the first 84 days (12 weeks) of the study (28 days, or 4 weeks for Cohort 1):

  * Shares a household with a child <3 years of age, a pregnant woman or a woman who plans to become pregnant during this time;
  * Household or sexual contact with someone who has weakened immunity (such as someone with HIV infection, someone receiving treatment for cancer, or an elderly person > 70 yrs);
  * Occupation as a food-handler, childcare (for children <3 years), or health care worker with direct patient contact.
* A clinically significant abnormality on physical examination
* Results of blood tests as defined by protocol
* Positive pregnancy test during medical screening or within 24 hours of inoculation or current breast feeding (women).
* Failure to attain a score of at least 70% on the written examination (two attempts permitted)
* During the past 3 years, developed diarrhea during travel to a developing country, or within 1 week of returning home.
* Receipt of any of the following:

  * Any vaccine or investigational drug within 30 days of study vaccine
  * A live, attenuated vaccine within 30 days of the study vaccine
  * A subunit or killed vaccine within 14 days of the study vaccine
  * A blood product in the 90 days before the study vaccine
* Receipt of antibiotics within 7 days of inoculation (or within 21 days if the antibiotic was azithromycin).
* Loose stools or any other acute illness such as fever >100.0 degrees F during the 48 hours before vaccination.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with reactions and adverse events | Reactions are evaluated for 7 days after each dose. Adverse events are evaluated for the entire study participation (6 months for cohort 1 and 8 months for all other cohorts).
  occurence of diarrhea, dysentery and fever.
Number of participants who receive the vaccine who get immunity to shigella | Immunity in the blood will be assessed using serial samples collected during the 84 days after the first vaccination. Immunity at the intestinal level will be assessed by collecting seral stool samples for 14 days after each vaccination.
  It is hoped that the vaccine will trigger the body's immune system to make specific responses such as antibodies (special proteins) and antibody-producing cells that are believed to protect against illness if a person is exposed to certain illness-causing Shigella in the future.

SECONDARY OUTCOMES:
Number of participants who pass the vaccine in their stool | The first 84 days after vaccination
  Volunteers' stool will be tested to see if the vaccine is present. This will tell whether the vaccine is able to stick to the intestine and grow there. We will see whether this information predicts the strength of the immune responses to the vaccine and whether the vaccine could potentially be passed to close contacts.
The number of participants who develop various types of immune responses | The first 84 days of the study
  We will look at the ability of the vaccine to evoke different types of responses in blood and stool that might protect them against Shigella infections in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Karen L. Kotloff, M.D., Principal Investigator — University of Maryland,Baltimore Center for Vaccine Development
Locations (2):
- United States (2):
  - Shin Nippon Biomedical Laboratories, LTD. (SNBL) Inpatient Facility, Baltimore, Maryland
  - University of Maryland, Baltimore Center for Vaccine Development, Baltimore, Maryland

REFERENCES:
- [Derived] Toapanta FR, Bernal PJ, Kotloff KL, Levine MM, Sztein MB. T cell mediated immunity induced by the live-attenuated Shigella flexneri 2a vaccine candidate CVD 1208S in humans. J Transl Med. 2018 Mar 13;16(1):61. doi: 10.1186/s12967-018-1439-1. PMID 29534721